CLINICAL TRIAL: NCT04422132
Title: Randomized Phase II Trial of Salvage Radiotherapy for Prostate Cancer In 4 Weeks v. 2 Weeks
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Viewray Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-03021572
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ARM 1 - 2 weeks (Active Comparator): Patients will receive treatment to the prostate fossa +/- nodes in 32.5 Gy in 5 fractions. Patients receiving 32.5 Gy in 5 fractions cannot be treated on consecutive days.
  Interventions: Radiation: 5 days Radiation Therapy (32.5 Gy in 5 fractions)
- ARM 2 - 4 weeks (Active Comparator): Patients will receive treatment to the prostate fossa +/- nodes in 55 Gy in 20 fractions.
  Interventions: Radiation: 20 days Radiation therapy (55 Gy in 20 fractions)

INTERVENTIONS:
Radiation: 5 days Radiation Therapy (32.5 Gy in 5 fractions) — Patients will receive treatment to the prostate fossa +/- nodes in either 32.5 Gy in 5 fractions or 55 Gy in 20 fractions.
  Arms: ARM 1 - 2 weeks
Radiation: 20 days Radiation therapy (55 Gy in 20 fractions) — Patients will receive treatment to the prostate fossa +/- nodes in either 32.5 Gy in 5 fractions or 55 Gy in 20 fractions.
  Arms: ARM 2 - 4 weeks

SUMMARY:
The purpose of this study is to compare urinary and bowel side effects of hypofractionated radiotherapy in 20 treatments (4 weeks) to ultra-hypofractionated radiotherapy in 5 treatments (2 weeks) for prostate cancer that has returned after prostatectomy. The investigators are also interested in looking at time to progression and the quality of life (health scores).

DETAILED DESCRIPTION:
The standard treatment for most patients with biochemical recurrence after radical prostatectomy is salvage radiotherapy. Salvage radiotherapy delays the need for chronic, non-curative treatment, such as long-term androgen suppression, and is the only potentially curative treatment of some biochemical recurrences after prostatectomy.

Patients are recommended to undergo salvage radiotherapy to eradicate biochemical disease delivered in approximately 40 treatments over the course of 8 weeks, representing a high burden of therapy, which may be related to lower utilization of salvage radiotherapy. Modern radiotherapy for prostate cancer has been afforded many advantages including advanced image-guided radiotherapy allowing for larger dose delivery in fewer treatments and smaller margins with hypofractionated (20 treatments) and ultra-hypofractionated (5 treatments) radiotherapy.

In patients that need salvage radiotherapy, the potential advantages of hypofractionated and ultra-hypofractionated radiotherapy delivered over 20 or 5 treatments are: 1) increased convenience to patients because of fewer treatment days, 2) reduced costs to patients because of reduced travel expenses and copays, 3) improved resource utilization for physicians because of the fewer number of treatments per patient and consequently 4) reduced cost to society. In prostate cancer specifically, hypofractionated and ultra-hypofractionated radiotherapy has the added potential of not increasing toxicity with shorter treatment times.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 and older with histologically confirmed prostate cancer after prostatectomy with detectable PSA. PSA does not need to be detectable for men with pathologically node positive disease.
* KPS >=70
* Patient with no evidence of distant metastatic disease on PET/CT/MRI or bone scan < 9 months prior to enrollment. Patients with positive pelvic lymph nodes are eligible.
* Ability to receive MRI-guided radiotherapy.
* Equivocal evidence of metastatic disease outside the pelvis on standard imaging requires documented negative biopsy.
* Ability to complete the Expanded Prostate Cancer Index Composite (EPIC) questionnaire.

Exclusion Criteria:

* Prior history of receiving pelvic radiotherapy.
* Patient with inflammatory bowel disease.
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of ultra-hypofractionated radiotherapy.
* History of bladder neck or urethral stricture.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 134 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of patient-reported GI symptoms using the Expanded Prostate Cancer Index Composite (EPIC) | Baseline, 1 month, 24 months
  The primary objective is to demonstrate that 5 days of ultra-hypofractionated radiotherapy does not significantly increase patient-reported Gastrointestinal (GI) and Genitourinary (GU) symptoms over 20 days of hypofractionated radiotherapy 2 years after treatment completion as measured by EPIC.
  Expanded Prostate Cancer Index Composite (EPIC) short form questionnaire. The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. Scores range from 0 to 100, lower scores indicate worse outcomes and higher EPIC scores represent better outcomes.

SECONDARY OUTCOMES:
Change in the number of patient reported GI-GU symptoms at specific intervals as measured by Expanded Prostate Cancer Index Composite (EPIC) | 3 months, 6 months, 12 months, 24 months, 60 months
  Secondary endpoints will include both the safety endpoints including change in GI and GU symptoms at 3, 6, 12, 24 and 60 months from end of treatment as measured by EPIC.
  Expanded Prostate Cancer Index Composite (EPIC) short form questionnaire. The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. Scores range from 0 to 100, lower scores indicate worse outcomes and higher EPIC scores represent better outcomes.
  Adverse events can be unexpected or expected, related to treatment.
Time to progression (TTP) | 3 months, 6 months, 12 months, 24 months, 60 months
  Compare time to progression (TTP) where progression is defined as the first occurrence of biochemical failure (BF), local failure, regional failure, distant metastasis (DM), institution of new unplanned anticancer treatment, or death from prostate cancer (PCSM).
Overall survival (OS) | 3 months, 6 months, 12 months, 24 months, 60 months
  Overall survival (OS) will be measured among the participants
Number of patients who expired due to prostate cancer. | Through study completion, an average of 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Emily Weg, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marciscano AE, Wolfe S, Zhou XK, Barbieri CE, Formenti SC, Hu JC, Molina AM, Nanus DM, Nauseef JT, Scherr DS, Sternberg CN, Tagawa ST, Nagar H. Randomized phase II trial of MRI-guided salvage radiotherapy for prostate cancer in 4 weeks versus 2 weeks (SHORTER). BMC Cancer. 2023 Aug 22;23(1):781. doi: 10.1186/s12885-023-11278-3. PMID 37608258
- See also: Related Info — https://expl.ai/JUCWKDB